CLINICAL TRIAL: NCT06044935
Title: Effect of Nicotinamide Riboside on Ketosis, Fat Oxidation &Amp;Amp;Amp;Amp; Metabolic Rate
Brief Title: Effect of Nicotinamide Riboside on Ketosis, Fat Oxidation & Metabolic Rate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 10001690; 001690-DK
Record Dates: First submitted 2023-09-19; First posted 2023-09-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Overweight; Obesity
Keywords: Ketogenic Diet; Sleep; Energy Expenditure; Supplement; Calories
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet, Ketogenic; nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Men with overweight or obesity (Experimental): To investigate whether NR supplementation augments the sleeping energy expenditure and fat oxidation rate during the ketogenic diet in men and women with overweight and obesity
  Interventions: Other: Standard Diet; Other: Ketogenic Diet; Dietary Supplement: Placebo; Dietary Supplement: Nicotinamide Riboside
- MODY2 Patients (Experimental): To measure changes in sleeping energy expenditure and fat oxidation rate after transitioning from a baseline diet to an isocaloric ketogenic diet similar to our previous study in men
  Interventions: Other: Standard Diet; Other: Ketogenic Diet; Dietary Supplement: Placebo
- Women with overweight or obesity (Experimental): To investigate whether NR supplementation augments the sleeping energy expenditure and fat oxidation rate during the ketogenic diet in men and women with overweight and obesity
  Interventions: Other: Standard Diet; Other: Ketogenic Diet; Dietary Supplement: Placebo; Dietary Supplement: Nicotinamide Riboside

INTERVENTIONS:
Other: Standard Diet — Consisting of 15% protein, 35% fat, and 50% carbohydrate, matching the macronutrient composition of a typical American diet
Other: Ketogenic Diet — Consisting of a macronutrient composition of 15% protein, 80% fat, and 5% carbohydrate
Dietary Supplement: Placebo — Subjects without MODY2 will take either placebo or NR (1 g BID, 2 g per day total) supplements for 7 days during this Run-in phase
Dietary Supplement: Nicotinamide Riboside — Subjects without MODY2 will take either placebo or NR (1 g BID, 2 g per day total) supplements for 7 days during this Run-in phase
  Arms: Men with overweight or obesity; Women with overweight or obesity

SUMMARY:
Background:

At least 30% of Americans have fatty liver disease. This means that they store too much fat in the liver. At the moment lifestyle changes are the only way to treat this problem.

Objective:

To test how (1) a low-carbohydrate diet and (2) a supplement called nicotinamide riboside (NR) affect how a person s body uses dietary fat.

Eligibility:

Men aged 18 to 65 and women aged 18 to 50 who are healthy volunteers with a body mass index (height to weight ratio) of 25 or more. Adults with maturity-onset diabetes of the young type 2 (MODY2) are also needed.

Design:

Participants with diabetes will have 1 screening visit and a 9-day clinic stay. Healthy volunteers will have 1 screening visit and 2 clinic stays of 1 to 2 weeks each.

During screening, all participants will have a physical exam with blood and urine tests. They will have their heart rhythm measured while riding a gym bike.

NR is a pill taken by mouth. Only healthy volunteers will take the NR, for 14 days at a time, during 1 clinic stay. During their other stay, they will take placebos; these are pills that look like the study supplement but contain no NR.

During each clinic stay, all participants will eat a normal American diet. Then they will eat a ketogenic "low-carb" diet for 5 days.

Participants will have many tests, including:

Sleeping every night and having two 24-hour stays in a special room that measures the gases their body uses and produces.

Drinking a high-fat shake, then remaining seated for 5 hours while their blood and breath are monitored.

Having a substance injected into the arm and remaining seated for 3 hours while their blood is measured.

Wearing monitors to measure their activity levels. Another monitor will measure their blood glucose levels.

Having imaging scans.

...

DETAILED DESCRIPTION:
Study Description:

This is a randomized, double-blind, placebo-controlled crossover study of adults with overweight or obesity to determine whether nicotinamide riboside supplementation increases sleeping energy expenditure and fat oxidation rate during a ketogenic diet.

Objectives:

Primary Aim 1: Determine whether sleeping energy expenditure increases after transitioning to a low carbohydrate ketogenic diet as compared to a baseline high carbohydrate run-in diet in men

Primary Aim 2: Determine whether sleeping energy expenditure is affected by NR supplementation during a ketogenic diet in men

Secondary Aim 1: Determine whether fat oxidation during sleep increases after transitioning to a low carbohydrate ketogenic diet as compared to a baseline high carbohydrate run-in diet in men

Secondary Aim 2: Determine whether fat oxidation during sleep is affected by NR supplementation during a ketogenic diet from the baseline run-in diet in men

Exploratory Aims: Exploratory comparison of the above endpoints between men and women without MODY2.

Exploratory comparison of the above diet-related endpoints between patients with MODY2 and those obtained during the Placebo period in other participants.

Several exploratory measurements are planned to help comprehensively phenotype the effects of the diets and nicotinamide riboside supplementation and are intended to be hypothesis-generating. We will assess the following:

* Liver TG
* Daily ketosis, insulin secretion, and protein utilization
* Rates of ketogenesis and lipolysis
* Physical activity and sleep assessment
* Body composition assessment
* Fasting and postprandial blood measurements of various metabolites, hormones, cytokines, and markers of inflammation.
* Microbiome composition
* Hunger and satiety before and after meals
* Eating rate
* Chronotype and sleep quality
* Usual food intake
* 24-h and exercise energy expenditure

Endpoints:

Primary:

Mean change in sleeping energy expenditure between the ketogenic diet and the baseline run-in diet

Mean difference in sleeping energy expenditure between NR and placebo during the ketogenic diet

Secondary:

Mean change in sleeping fat oxidation rate between the ketogenic diet and the baseline run-in diet Mean difference in fat oxidation rate between NR and placebo during the ketogenic diet

Exploratory:

* H magnetic resonance spectroscopy
* 24hr urine ketones, C-peptide, nitrogen
* Stable isotope infusions of 13C beta-hydroxybutyrate and 2H glycerol
* Daily accelerometry and wireless EEG headband
* DXA scans
* Fasting and postprandial blood concentrations of various metabolites, hormones, cytokines and inflammatory markers
* Blood glucose variability and mean concentration as measured by Continuous Glucose Monitoring
* Daily fasting glucose and beta-hydroxybutyrate concentrations by finger-prick
* Microbiome composition
* Hunger and satiety visual analogue scores
* Meal duration
* Pittsburg sleep quality index, morningness-eveningness questionnaire, and subjective sleep visual analogue scores
* Usual food intake as measured by Food frequency questionnaire
* 24-h and exercise energy expenditure from metabolic chamber

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Meet one of the following:

   1. Adult males aged 18-65 years
   2. Pre-menopausal adult females aged 18-50 years
   3. Adult males aged 18-65 years with diagnosed maturity-onset diabetes of the young type 2 (MODY2) or pre-menopausal adult females aged 18-50 years with diagnosed MODY2
2. Weight stable (< +/- 5 % body weight change over past 6 months) as determined by volunteer report
3. Body mass index (BMI) >= 25 kg/m^2 (of >=18.5 kg/m^2 for patients with MODY2)
4. Able to cycle at a moderate rate and intensity with a HR equal to or greater than 0.3x(220-age-HRrest)+HRrest but not exceeding 0.4x(220-age-HRrest)+HRrest with no signs of arrhythmia

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Taking prescription medications or other drugs or supplements that may influence energy metabolism or nutrient digestion or absorption (including, but not limited to, diet/weight-loss medication or other medications at the discretion of the PI and/or study team)
2. Indicators of liver disease; combination of both albumin < 2.8 mg/mL and bilirubin > 3 mg/mL
3. Individuals with significant medical comorbidities (e.g., non-MODY2 diabetes, NYHA Class >II heart failure, or CKD Stage II or worse, or American Society of Anesthesiologists Physical Status Class 3 or above)
4. Individuals taking prescription medications to treat hypertension in participants without MODY2
5. Participating in a regular exercise program (> 2h/week of vigorous activity) as determined by volunteer report
6. Positive pregnancy test (only for people who can get pregnant)
7. Hematocrit < 40% (men only)
8. Hematocrit <37% (women only)
9. Caffeine consumption > 300 mg/day as determined by volunteer report
10. Alcohol consumption > 3 drinks per day for men or > 2 drinks per day for women as determined by volunteer report
11. Regular use of tobacco (smoking or chewing), e-cigarettes (a.k.a. vapes), nicotine patches, or illicit drugs over past 6 months as determined by volunteer report. Subjects may also be excluded based on a urine drug test.
12. Psychological conditions as determined by volunteer report such as (but not limited to) eating disorders, depression, bipolar disorders, that would be incompatible with safe and successful participation in this study, as determined by investigators
13. Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, food allergies) or a reported dislike of a significant fraction of the study foods
14. Unwilling or unable to comply with or perform all study procedures (e.g. cycling or activities of daily living), or unavailability for the duration of the study, as determined by participant or investigator discretion
15. Unwilling or unable to adhere to Lifestyle Considerations throughout study duration, as determined by participant or investigator discretion
16. Volunteers unwilling or unable to give informed consent
17. Participants with a measured Resting Energy Expenditure (REE) more than 30% above or below the predicted REE based on Mifflin St Jeor equation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in sleeping energy expenditure between the ketogenic diet and the baseline run-in diet | 7 days
  Mean change in sleeping energy expenditure measured by room calorimetry from 2 days of standard run-in diet to 5 days of ketogenic diet
Mean difference in sleeping energy expenditure between NR and placebo during the ketogenic diet | 5 days
  Mean difference in sleeping energy expenditure measured by room calorimetry during 5 days of ketogenic diet with NR supplementation or placebo

SECONDARY OUTCOMES:
Mean change in sleeping fat oxidation rate between the ketogenic diet and the baseline run-in diet | 7 days
  Mean change in sleeping fat oxidation measured by room calorimetry from 2 days of standard run-in diet to 5 days of ketogenic diet
Mean difference in fat oxidation rate between NR and placebo during the ketogenic diet | 5 days
  Mean difference in sleeping fat oxidation measured by room calorimetry during 5 days of ketogenic diet with NR supplementation or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Chung, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
demographics, anthropometrics, indirect calorimetry data, circulating metabolites and hormones
Supporting Information: Study Protocol, Analytic Code
Time Frame: Upon publication in peer reviewed journal
Access Criteria: Open

REFERENCES:
- [Background] Hall KD, Chen KY, Guo J, Lam YY, Leibel RL, Mayer LE, Reitman ML, Rosenbaum M, Smith SR, Walsh BT, Ravussin E. Energy expenditure and body composition changes after an isocaloric ketogenic diet in overweight and obese men. Am J Clin Nutr. 2016 Aug;104(2):324-33. doi: 10.3945/ajcn.116.133561. Epub 2016 Jul 6. PMID 27385608
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001690-DK.html